CLINICAL TRIAL: NCT06898229
Title: Effect of Audiovisual Education on Breast Cancer Screening and Fear in Illiterate Women
Brief Title: Effect of Audiovisual Education on Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Nurten Terkes, Principal Investigator, Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GO 2022/857
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Educational Status

STUDY DESIGN:
Masking Description: They did not know if they were in the control and intervention group at the time of randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Active Comparator): It focussed on informing and raising awareness. In this process, basic information about the definition, importance, risk factors and symptoms of breast cancer was conveyed through audio-visual materials supported by short videos, animations and photographs. In addition, group discussions were organised on the importance of breast cancer screening, the advantages of early diagnosis, and fears and concerns about breast cancer. At the end of the training, the simulation applications were evaluated and the questions and concerns of the participants were discussed. The trainings were repeated at the first follow-up, 3rd month and 6th month and the long-term effects of the study were evaluated.
  Interventions: Behavioral: Education
- Control (No Intervention): Participants in the control group did not receive any treatment.

INTERVENTIONS:
Behavioral: Education — The intervention program aimed to increase participation in breast cancer screenings and reduce fear among illiterate women. The three-month training was structured in three phases. In the first month, awareness was raised through visual-audio materials about breast cancer, risk factors, and the importance of early diagnosis. In the second month, practical training was provided on breast self-examination (BSE), and clinical breast examination (CBE) and mammography procedures were introduced. In the final month, group discussions and success stories supported behavioral change, reinforcing knowledge. The program's effectiveness was evaluated through pre-test and post-test comparisons.
  Arms: Education

SUMMARY:
This study was conducted as a double-blind randomised controlled trial to determine the effect of education using audio-visual methods and simulation techniques on breast cancer screening and breast cancer fears in illiterate women. The study was conducted in the villages of a district in the south of Turkey with a distance of over 100 km to health institutions. The sample size of the study was calculated with the G*Power 3.1 programme based on the mean breast cancer fear scores (22.42±8.30 for those without family history and 28.14±6.23 for those with family history) in a study, with a 95% confidence interval, 5% margin of error, 0.92 effect size and 95% power. As a result of this analysis, the minimum sample size required was determined as 64 people in total. However, a total of 120 women were included in the study in order to increase the power of the research, to prevent possible data loss and to make the results more reliable. Participants were divided into intervention (n=60) and control (n=60) groups by simple random sampling method.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 40-69 (Republic of Turkey Ministry of Health, 2020a).
2. Being a woman living in rural areas.
3. Being an illiterate woman.
4. Not being diagnosed with breast cancer.
5. Not being pregnant, breastfeeding or puerperant.
6. Accepting to participate in the study.
7. Absence of a mental illness.
8. No communication barriers

Exclusion Criteria:

1. Not having completed the given training sessions
2. Having had problems with breast cancer before.
3. Having breast conserving surgery for any reason.

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Illiterate Women
Enrollment: 160 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Champion Breast Cancer Fear Scale | 5-10 minutes
  The Scale is an 8-item measurement tool developed by Victoria Champion et al. in 2004. In the original study of the scale, Cronbach's alpha coefficient was found to be 0.91 for African-American and white women and 0.94 for African-American women. This scale was developed to determine the relationship between breast cancer, mammography behaviour and women's emotional reactions and is a Likert-type scale scored from 1 to 5. The highest score to be obtained from the scale is 40 and the lowest score is 8. In the evaluation of the scores; 8-15 points indicate low level fear, 16-23 points indicate medium level fear and 24-40 points indicate high level fear. Breast Cancer Fear Scale was adapted into Turkish by Seçginli in 2012.

SECONDARY OUTCOMES:
Post-Training Screening Behaviour Follow-up Form | 5-10 minutes
  This form was used as a post-test after the training and follow-up of the women. With this form, it was determined which of the early diagnosis practices such as CHC, MMC and mammography the women performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Burdur Mehmet Akif Ersoy University, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
All authors contributed to the interpretation, writing, and approval of the final manuscript.

REFERENCES:
- [Result] Ozdemir A, Unal E. The effect of breast self-examination training on nursing students by using hybrid-based simulation on knowledge, skills, and ability to correctly evaluate pathological findings: Randomized Controlled Study. Nurse Educ Pract. 2023 Jan;66:103530. doi: 10.1016/j.nepr.2022.103530. Epub 2022 Nov 29. PMID 36462274
- [Result] Joulaei H, Delshad MH, Pourhaji F. The Correlation of Social Support and Fear of Breast Cancer among Women in Northeast of Iran: A Cross-Sectional Study. Int J Community Based Nurs Midwifery. 2023 Jul;11(3):210-221. doi: 10.30476/IJCBNM.2023.98094.2225. PMID 37489226
- [Result] Champion VL, Skinner CS, Menon U, Rawl S, Giesler RB, Monahan P, Daggy J. A breast cancer fear scale: psychometric development. J Health Psychol. 2004 Nov;9(6):753-62. doi: 10.1177/1359105304045383. PMID 15367754